CLINICAL TRIAL: NCT02268110
Title: The Effect of Exercise Therapy and/or Abdominal Binding on Inter-rectus Distance, Abdominal Muscle Strength, Lumbopelvic and Urogynecological Complaints, Perceived Function, and Body Image in Post-partum Women With Diastasis Recti
Brief Title: The Effect of Conservative Interventions on the Signs and Symptoms of Diastasis Recti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Nadia Keshwani, PhD candidate, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REH-566-13
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Diastasis Recti And Weakness Of The Linea Alba
Keywords: diastasis recti; physiotherapy; exercise therapy; abdominal binding
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Supervised exercise therapy (Experimental): Participants will receive 12 sessions with a physiotherapist where they will receive instructions on body mechanics, and be given a progressive abdominal exercise program
  Interventions: Other: Exercise therapy
- Abdominal binding (Experimental): Participants will be fitted for an abdominal binder and asked to wear it for a period of 12 weeks.
  Interventions: Other: Abdominal binding
- Exercise therapy and Abdominal Binding (Experimental): Participants will attend 12 sessions with a physiotherapist, and receive an abdominal binder
  Interventions: Other: Exercise therapy; Other: Abdominal binding
- Control (No Intervention): Participants will not receive an intervention during the study period

INTERVENTIONS:
Other: Exercise therapy — Supervised exercise therapy with a 12 week progressive abdominal exercise home program for
  Arms: Exercise therapy and Abdominal Binding; Supervised exercise therapy
Other: Abdominal binding — Wearing an abdominal binder for 12 weeks
  Arms: Abdominal binding; Exercise therapy and Abdominal Binding

SUMMARY:
The purpose of this study is to determine the effect of two different physiotherapeutic interventions (exercise therapy and/or abdominal binding) on the signs and symptoms of diastasis recti in post-partum women.

DETAILED DESCRIPTION:
This study is investigating the effect of exercise therapy and/or abdominal binding on inter-rectus distance, abdominal muscle strength and endurance, lumbopelvic dysfunction, urogynecological complaints, perceived function, and body image in post-partum women with diastasis recti

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years old
* given birth to their first child, vaginally, in the last three to four weeks
* inter-rectus distance of two finger widths of greater on palpation during head lift

Exclusion Criteria:

* history of persistent pain with intercourse prior to pregnancy
* diagnosed with neurological impairments affecting the central nervous system or sacral nerves
* diagnosed with connective tissue disorders

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-08; Primary Completion 2017-08 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Inter-Rectus Distance | baseline, 12 weeks post intervention, 9 months post intervention
  Measured using ultrasound imaging

SECONDARY OUTCOMES:
Change in Abdominal Strength and Endurance | baseline, 12 weeks post intervention, 9 months post intervention
  measured using clinical tests and hand-held dynamometry
Change in Body image | baseline, 12 weeks post intervention, 9 months post intervention
  measured using the Multidimensional Body-Self Relations Questionnaire
Change in Lumbopelvic dysfunction | baseline, 12 weeks post intervention, 9 months post intervention
  measured using Modified Oswestry Questionnaire
Change in Urogynecological Complaints | baseline, 12 weeks post intervention, 9 months post intervention
  measured using the Pelvic Floor Distress Inventory
Change in Severity of Lumbopelvic and/or Abdominal Pain | baseline, 12 weeks post intervention, 9 months post intervention
  Visual Analog Scale
Change in Perceived Function | baseline, 12 weeks post intervention, 9 months post intervention
  Inventory of Functional Status After Childbirth Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: McLean Linda, PhD, Study Director — Queen's University
Locations (1):
- Rehabilitation Sciences Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No